CLINICAL TRIAL: NCT02802241
Title: Effects of Open-label vs Double-blind Treatment in IBS.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Judy Nee, Assistant Professor of Medicine, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Purpose: Treatment
Other Study IDs: 2015P000282; R01AT008573 (NIH)
Record Dates: First submitted 2016-06-14; First posted 2016-06-16 (Estimated); Results first posted 2020-09-04 (Actual); Last update posted 2024-01-22 (Actual); Status verified 2024-01

CONDITIONS: Irritable Bowel Syndrome; Placebo Effect; Placebos; Peppermint Oil
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — peppermint oil

ARMS (4):
- open-label placebo (Experimental)
  Interventions: Drug: placebo
- double-blind placebo (Experimental)
  Interventions: Drug: placebo
- double-blind peppermint oil (Experimental)
  Interventions: Dietary Supplement: peppermint oil
- no additional treatment (No Intervention)

INTERVENTIONS:
Drug: placebo
  Arms: double-blind placebo; open-label placebo
Dietary Supplement: peppermint oil
  Arms: double-blind peppermint oil

SUMMARY:
The purpose of this study is to investigate placebo effects and peppermint oil in Irritable Bowel Syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Meet Rome IV diagnostic criteria for IBS

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 340 (Actual)
Dates: Start 2016-06; Primary Completion 2019-01 (Actual); Study Completion 2019-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Lembo A, Kelley JM, Nee J, Ballou S, Iturrino J, Cheng V, Rangan V, Katon J, Hirsch W, Kirsch I, Hall K, Davis RB, Kaptchuk TJ. Open-label placebo vs double-blind placebo for irritable bowel syndrome: a randomized clinical trial. Pain. 2021 Sep 1;162(9):2428-2435. doi: 10.1097/j.pain.0000000000002234. PMID 33605656
- [Derived] Ballou S, Kaptchuk TJ, Hirsch W, Nee J, Iturrino J, Hall KT, Kelley JM, Cheng V, Kirsch I, Jacobson E, Conboy L, Lembo A, Davis RB. Open-label versus double-blind placebo treatment in irritable bowel syndrome: study protocol for a randomized controlled trial. Trials. 2017 May 25;18(1):234. doi: 10.1186/s13063-017-1964-x. PMID 28545508

RESULTS

PARTICIPANT FLOW:
Groups:
- Open-label Placebo; Double-blind Placebo: placebo
- Double-blind Peppermint Oil: peppermint oil
- no Pill Control: control
Period: Overall Study
Arm/Group | Open-label Placebo | Double-blind Placebo | Double-blind Peppermint Oil | no Pill Control
Started (intention to treat) | 89 | 87 | 46 | 86
Planned Analysis | 89 | 87 | 46 (Not included in primary analysis) | 86
Completed | 68 | 71 | 30 (Not included in primary analysis) | 72
Not Completed | 21 | 16 | 16 | 14

BASELINE CHARACTERISTICS:
Population: Intention to treat. Double-blind peppermint oil was not collected in the intention to treat.
Groups:
- Total: Total of all reporting groups
Arm/Group | Open-label Placebo | Double-blind Placebo | no Pill Control | Double-blind Peppermint Oil | Total
Number analyzed (Participants) | 89 | 87 | 86 | 46 | 308
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.2 (17.6) | 43.8 (19.2) | 40.0 (17.7) | 41.0 (17.4) | 42.0 (18.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 63 | 64 | 63 | 34 | 224
  Male | 26 | 23 | 23 | 12 | 84
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 3 | 4 | 9 | 2 | 18
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 4 | 3 | 5 | 3 | 15
  White | 73 | 75 | 66 | 41 | 255
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 9 | 5 | 6 | 0 | 20
IBS-SSS [Mean (Standard Deviation); unit: units on a scale] | 286.0 (62) | 285.8 (69.0) | 274.4 (71.1) | 283.5 (71.7) | 282.1 (67.4)

OUTCOME MEASURES:

1. Primary Outcome: Change in Irritable Bowel Syndrome - Symptom Severity Score (IBS-SSS) From Baseline to Six Weeks.
Description: Score ranges from 0-500, 0 indicates no symptoms, 500 indicates worst possible symptoms
Time Frame: 6 weeks
Population: Double-blind peppermint oil data was not part of the planned analysis. While the data was collected, the results were analyzed with a modified intention to treat which differs from the primary analysis of intention to treat. The outcome results data are not an accurate comparision.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Open-label Placebo | Double-blind Placebo | no Pill Control | Double-blind Peppermint Oil
Number analyzed (Participants) | 89 | 87 | 86 | 46
score on a scale
  intention to treat | 74.6 [47.3 to 101.8] | 94.6 [71.8 to 117.4] | 56.4 [31.4 to 81.4] | 90.8 [45 to 102]
  planned analysis | 90.6 [68.6 to 112.6] | 100.3 [78.7 to 121.8] | 52.3 [30.8 to 73.7] | 90.8 [75.3 to 110]

ADVERSE EVENTS:
Time Frame: 6 weeks
Description: Participants are not at risk for adverse events or mortality since they were not given an active medication. Double-blind peppermint oil data was not collected as part of this study.
Arm/Group | Open-label Placebo | Double-blind Placebo | Double-blind Peppermint Oil | no Pill Control
All-Cause Mortality (participants affected / at risk) | 0/96 | 0/97 | 0/0 | 0/98
Serious Adverse Events (participants affected / at risk) | 0/96 | 0/97 | 0/0 | 0/98
Other Adverse Events (participants affected / at risk) | 5/96 | 11/97 | 0/0 | 0/98
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open-label Placebo (N=96) | Double-blind Placebo (N=97) | Double-blind Peppermint Oil (N=0) | no Pill Control (N=98)
diarrhea (Gastrointestinal disorders) | 5 (5) | 5 (5) | 0 (0) | 0 (0)
heartburn (Gastrointestinal disorders) | 1 (1) | 6 (6) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-06-15): https://cdn.clinicaltrials.gov/large-docs/41/NCT02802241/Prot_SAP_001.pdf
  • Informed Consent Form (2018-08-17): https://cdn.clinicaltrials.gov/large-docs/41/NCT02802241/ICF_000.pdf